CLINICAL TRIAL: NCT05167747
Title: Double-blind, Placebo-controlled, Randomized Clinical Trial Comparing the Effect of a Combined Nutraceutical and Placebo on Blood Pressure Level, Vascular Health, and Metabolic Parameters in Subjects Affected by Normal-High Blood Pressure
Brief Title: Food Supplementation With Diuripres for Blood Pressure Modulation in Subjects With High-Normal Blood Pressure
Acronym: CONDOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Arrigo F.G. Cicero, Prof., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pre-HPT_RCT_2021
Record Dates: First submitted 2021-05-28; First posted 2021-12-22 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: High-Normal Blood Pressure
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Dietary supplement
  Interventions: Dietary Supplement: Dietary Supplement
- Placebo comparator (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — Dietary supplement formulated with magnesium, standardized extract of orthosiphon, standardized extract of hawthorn and standardized extract of hibiscus. Each tablet contains: 0.1 g magnesium, 0.25 g standardized extract of orthosiphon (Orthosiphon stamineus Benth), 0.16 standardized extract of hawthorn (Crataegus curvisepala Lind.) and 0.08 g standardized extract of hibiscus (Hibiscus sabdariffa L.).
  Oral administration: 2 tablets/day at evening meal
  Arms: Active Comparator
Other: Placebo — Oral administration: 2 tablets/day at evening meal
  Arms: Placebo comparator

SUMMARY:
Cardiovascular diseases (CVDs) are the leading cause of mortality worldwide, reaching the 31% of deaths in 2012. CVDs represent also the major cause of disability in developed countries and has been estimated that their growing burden could lead to a global increase in loss of disability-adjusted life years (DALY), from a loss of 85 million DALYs of 1990 to a loss of ~ 150 million DALYs in 2020, becoming a major cause of no psychic responsible for lost productivity.

Several risk factors contribute to the aetiology and development of CVD. These factors have been traditionally stratified into modifiable risk factors through the lifestyle changes or by taking a pharmacologic treatment (e.g. hypertension, smoking, diabetes mellitus, hypercholesterolemia) and not modifiable risk factors (age, male sex and family history). Essential hypertension is the most common modifiable risk factor in the general population, with a prevalence in Western Countries -including Italy- ranging between about 25-45%.

Given the large prevalence of the disease of the general population, hypertension is responsible for the vast majority of CVD in individuals with different CV risk profiles, despite the availability of effective and well tolerated antihypertensive therapies. In this regard, several reports have shown that hypertensive patients often present additional CV and metabolic risk factors, mostly hypercholesterolemia, hypertriglyceridemia, metabolic syndrome and diabetes, which further contribute to increase the individual risk of developing hypertension-related complications, including stroke, end-stage renal disease, congestive heart failure, and CVD death. The concomitant presence of hypertension and dyslipidaemia is also responsible for the objective difficulty in achieving the recommended therapeutic targets for BP and cholesterol levels in a setting of clinical practice.

Several pharmacological and non-pharmacological interventions have been proposed for ameliorating the relatively low rates of control of hypertension. Among these, an extensive use of nutrients and food supplements has been shown to provide favourable effects in the management and control of high-normal blood pressure (BP) (or pre-hypertension), that increases the risk of developing hypertension, cardiovascular diseases, and renal failure.

DETAILED DESCRIPTION:
Among food supplements largely used in this field, Orthosiphon stamineus Benth leaf extract has been recognized for its well-known diuretic properties; extract of hawthorn (Crataegus curvisepala Lind.) has been shown to exert a renal-protective effect in high salt-induced hypertension and extract of hibiscus (Hibiscus sabdariffa L.) is well known for its antihypertensive and vasodilator effect in human. Moreover, supplementation with magnesium has been recently found to play a critical role in BP regulation, through directly stimulating prostacyclin and nitric oxide formation, modulating endothelium-dependent and endothelium-independent vasodilation, reducing vascular tone and reactivity, and preventing vascular injury via its antioxidant and anti-inflammatory functions.

The objective of this study is to evaluate the effect of dietary supplementation of a combined food supplement (NUT) containing magnesium, standardized extract of orthosiphon (Orthosiphon stamineus Benth), standardized extract of hawthorn (Crataegus curvisepala Lind.) and standardized extract of hibiscus (Hibiscus sabdariffa L.) compared to placebo, on blood pressure and other markers of vascular aging in subjects with high-normal blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects agree to participate in the study and having dated and signed the informed consent form;
* Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements;
* Subjects with high-normal blood pressure (SBP= 130-139 mmHg and/or DBP= 85-89 mmHg);
* Subjects who, according to the SCORE charts, have a low or moderate cardiovascular risk (defined as a total cardiovascular risk < 5%) and for whom, according to 2018 ESC/ESH guidelines, the intervention strategy does not require a pharmacological intervention.

Exclusion Criteria:

* Subjects already affected by cardiovascular diseases (secondary prevention) or with an estimated 10 years cardiovascular disease risk> 5%;
* Obesity (Body mass index>30 kg/m2);
* Type 1 or type 2 diabetes;
* Assumption of anti-hypertensive drugs or food supplements, or drugs potentially affecting blood pressure;
* Lipid-lowering treatment not stabilized since at least 2 months;
* Anticoagulants therapy;
* Known current thyroid, gastrointestinal or hepatobiliary diseases;
* Any medical or surgical condition that would limit the patient adhesion to the study protocol;
* Abuse of alcohol or drugs (current or previous);
* History of malignant neoplasia in the 5 years prior to enrolment in the study;
* History or clinical evidence of inflammatory disease such as severe arthritis, systemic lupus erythematosus or chronic inflammatory diseases or current therapy with immunosuppressive agents or long-term glucocorticoids;
* History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study;
* Known previous intolerance to one component of the tested nutraceuticals;
* Women in fertile age not using consolidated contraceptive methods;
* Pregnancy and Breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure absolute reduction from baseline and between groups | 8 weeks
  Absolute reduction of systolic blood pressure after 8 weeks of treatment
Diastolic blood pressure absolute reduction from baseline and between groups | 8 weeks
  Absolute reduction of diastolic blood pressure after 8 weeks of treatment

SECONDARY OUTCOMES:
Systolic blood pressure absolute reduction from baseline and between groups | 4 weeks
  Absolute reduction of systolic blood pressure after 4 weeks of treatment
Diastolic blood pressure absolute reduction from baseline and between groups | 4 weeks
  Absolute reduction of diastolic blood pressure after 4 weeks of treatment
Percent reduction from baseline and between groups in vascular reactivity | 4 weeks
  Percent reduction of flow-mediated dilation (FMD) after 4 weeks of treatment
Percent reduction from baseline and between groups in vascular reactivity | 8 weeks
  Percent reduction of flow-mediated dilation (FMD) after 8 weeks of treatment
Absolute change from baseline and between groups in body weight | 4 weeks
  Absolute change of body weight after 4 weeks of treatment
Absolute change from baseline and between groups in body weight | 8 weeks
  Absolute change of body weight after 8 weeks of treatment
Absolute change from baseline and between groups in body mass index | 4 weeks
  Absolute change of body mass index after 4 weeks of treatment
Absolute change from baseline and between groups in body mass index | 8 weeks
  Absolute change of body mass index after 8 weeks of treatment
Absolute change from baseline and between groups in waist circumference | 4 weeks
  Absolute change of waist circumference after 4 weeks of treatment
Absolute change from baseline and between groups in waist circumference | 8 weeks
  Absolute change of waist circumference after 8 weeks of treatment
Absolute change from baseline and between groups in hip circumference | 4 weeks
  Absolute change of hip circumference after 4 weeks of treatment
Absolute change from baseline and between groups in hip circumference | 8 weeks
  Absolute change of hip circumference after 8 weeks of treatment
Absolute change from baseline and between groups in waist/hip circumference ratio | 4 weeks
  Absolute change waist/hip circumference ratio after 4 weeks of treatment
Absolute change from baseline and between groups in waist/hip circumference ratio | 8 weeks
  Absolute change waist/hip circumference ratio after 8 weeks of treatment
Absolute change from baseline and between groups in the index of central obesity | 4 weeks
  Absolute change of the index of central obesity after 4 weeks of treatment
Absolute change from baseline and between groups in the index of central obesity | 8 weeks
  Absolute change of the index of central obesity after 8 weeks of treatment
Absolute change from baseline and between groups in the visceral adiposity index | 4 weeks
  Absolute change of the visceral adiposity index after 4 weeks of treatment
Absolute change from baseline and between groups in the visceral adiposity index | 8 weeks
  Absolute change of the visceral adiposity index after 8 weeks of treatment
Absolute change from baseline and between groups in fat and lean mass | 4 weeks
  Absolute change of fat and lean mass after 4 weeks of treatment
Absolute change from baseline and between groups in fat and lean mass | 8 weeks
  Absolute change of fat and lean mass after 8 weeks of treatment
Absolute change from baseline and between groups in renal function | 4 weeks
  Absolute change of creatinine and the estimated glomerular filtration rate (eGFR) after 4 weeks of treatment
Absolute change from baseline and between groups in renal function | 8 weeks
  Absolute change of creatinine and the estimated glomerular filtration rate (eGFR) after 8 weeks of treatment
Absolute change from baseline and between groups in serum lipids | 4 weeks
  Absolute change of serum concentrations of total cholesterol, triglycerides - TG, high-density lipoprotein cholesterol - HDL-C, non-high-density lipoprotein cholesterol - non HDL-C, low-density lipoprotein cholesterol - LDL-C after 4 weeks of treatment
Absolute change from baseline and between groups in lipids ratios | 4 weeks
  Absolute change of lipids ratios after 4 weeks of treatment
Absolute change from baseline and between groups in serum lipids | 8 weeks
  Absolute change of serum concentrations of total cholesterol, triglycerides - TG, high-density lipoprotein cholesterol - HDL-C, non-high-density lipoprotein cholesterol - non HDL-C, low-density lipoprotein cholesterol - LDL-C after 8 weeks of treatment
Absolute change from baseline and between groups in serum lipids ratios | 8 weeks
  Absolute change of lipids ratios after 8 weeks of treatment
Absolute change from baseline and between groups in high sensitivity C reactive protein | 4 weeks
  Absolute change of high sensitivity C reactive protein (hsCRP) after 4 weeks of treatment
Absolute change from baseline and between groups in high sensitivity C reactive protein | 8 weeks
  Absolute change of high sensitivity C reactive protein (hsCRP) after 8 weeks of treatment
Absolute change from baseline and between groups in serum uric acid concentrations | 4 weeks
  Absolute change of serum uric acid after 4 weeks of treatment
Absolute change from baseline and between groups in serum uric acid concentrations | 8 weeks
  Absolute change of serum uric acid after 8 weeks of treatment
Absolute change from baseline and between groups in fasting plasma glucose concentrations | 4 weeks
  Absolute change of fasting plasma glucose after 4 weeks of treatment
Absolute change from baseline and between groups in fasting plasma glucose concentrations | 8 weeks
  Absolute change of fasting plasma glucose after 8 weeks of treatment
Treatment acceptability | 4 weeks
  Evaluation of patients' satisfaction assessed by a Visual Analogue Scale (VAS) scale (with two end points representing 0 -low acceptability- and 10 -high acceptability-) after 4 weeks of treatment
Treatment acceptability | 8 weeks
  Evaluation of patients' satisfaction assessed by a Visual Analogue Scale (VAS) scale (with two end points representing 0 -low acceptability- and 10 -high acceptability-) after 8 weeks of treatment
Treatment tolerability | 4 weeks
  Evaluation of treatment's tolerability assessed by patients with a Visual Analogue Scale (VAS) scale (with two end points representing 0 -no pain- and 10 -pain as bad as it could possibly be-) after 4 weeks of treatment
Treatment tolerability | 8 weeks
  Evaluation of treatment's tolerability assessed by patients with a Visual Analogue Scale (VAS) scale (with two end points representing 0 -no pain- and 10 -pain as bad as it could possibly be-) after 8 weeks of treatment
Absolute change from baseline and between groups in liver transaminases and gamma glutamil transferase | 4 weeks
  Absolute reduction of alanine aminotransferase, aspartate aminotransferase and gamma glutamil transferase after 4 weeks of treatment
Absolute change from baseline and between groups in liver transaminases and gamma glutamil transferase | 8 weeks
  Absolute reduction of alanine aminotransferase, aspartate aminotransferase and gamma glutamil transferase after 8 weeks of treatment
Absolute change from baseline and between groups in augumentation pressure | 4 weeks
  Absolute change of augumentation pressure after 4 weeks of treatment assessed by Vicorder software
Absolute change from baseline and between groups in augumentation index | 4 weeks
  Absolute change of augumentation index after 4 weeks of treatment assessed by Vicorder software
Absolute change from baseline and between groups in augumentation pressure | 8 weeks
  Absolute change of augumentation pressure after 8 weeks of treatment assessed by Vicorder software
Absolute change from baseline and between groups in augumentation index | 8 weeks
  Absolute change of augumentation index after 8 weeks of treatment assessed by Vicorder software
Percent change from baseline and between groups in the estimated body water content | 4 weeks
  Percent change of the body water content after 4 weeks of treatment, assessed by bioelectrical impedance analysis (BIA)
Percent change from baseline and between groups in the estimated body water content | 8 weeks
  Percent change of the body water content after 8 weeks of treatment, assessed by bioelectrical impedance analysis (BIA)
Absolute change from baseline and between groups in estimated risk of cardiovascular disease | 4 weeks
  Absolute change of the percent estimated risk of cardiovascular disease after 4 weeks of treatment
Absolute change from baseline and between groups in estimated risk of cardiovascular disease | 8 weeks
  Absolute change of the percent estimated risk of cardiovascular disease after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arrigo F. Cicero, MD, Principal Investigator — S. Orsola-Malpighi University Hospital
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, Italy

REFERENCES:
- [Result] Fogacci F, Degli Esposti D, Di Micoli A, Fiorini G, Veronesi M, Borghi C, Cicero AFG. Effect of dietary supplementation with Diuripres(R) on blood pressure, vascular health, and metabolic parameters in individuals with high-normal blood pressure or stage I hypertension: The CONDOR randomized clinical study. Phytother Res. 2023 Oct;37(10):4851-4861. doi: 10.1002/ptr.7951. Epub 2023 Jul 14. PMID 37448322